CLINICAL TRIAL: NCT01608477
Title: Building Research Initiative Group: Chronic Illness Management and Adherence in Transplantation
Acronym: BRIGHT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Basel (Other)
Collaborators: KU Leuven (Other); University of Missouri, Kansas City (Other); Universitaire Ziekenhuizen KU Leuven (Other); Hospital Universitario À Coruña, Spain (Unknown); Azienda Ospedaliero, Universitaria Pisana (Other); Hannover Medical School (Other); Johns Hopkins University (Other); US Department of Veterans Affairs (U.S. Federal Agency); George Washington University (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Hopital Louis Pradel (Other); Hôpital Nord Laennec, France (Unknown); Groupe Hospitalier Pitie-Salpetriere (Other); University Hospital Heidelberg (Other); University Hospital, Udine, Italy (Other); University of Bologna (Other); Hospital de Sant Pau (Other); Puerta de Hierro University Hospital (Other); Hospital Universitario La Fe (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Zürich (Other); Papworth Hospital NHS Foundation Trust (Other Government); Freeman Hospital, UK (Unknown); Royal Brompton & Harefield NHS Foundation Trust (Other); Toronto General Hospital (Other); University of Ottawa Heart Institute, Canada (Unknown); St. Paul's Hospital, Canada (Other); London Health Sciences Centre (Other); Duke University Hospital, USA (Unknown); Virginia Commonwealth University (Other); The Cleveland Clinic (Other); Cedars-Sinai Medical Center (Other); Kaiser Permanente (Other); St Luke's Hospital, USA (Unknown); Hospital of the University of Pennsylvania, USA (Unknown); Ochsner Health System (Other); Hospital Israelita Albert Einstein (Other); Instituto Dante Pazzanese de Cardiologia (Other); Instituto do Coração da Universidade de São Paulo, Brazil (Unknown); St Vincent's Hospital, Sydney (Other); The Prince Charles Hospital (Other Government); Astellas Pharma Europe Ltd., UK (Unknown)
Responsible Party: Principal Investigator, Sabina De Geest, PhD, RN, FAAN, FRCN, University of Basel
Other Study IDs: BRIGHT
Record Dates: First submitted 2012-05-18; First posted 2012-05-31 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Heart Transplantation
Keywords: Heart transplantation; Medication adherence; Behavior system factor
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Over the past decades, survival rates in heart transplantation recipients improved significantly, due to advancements in regimens of immunosuppressives and surgical techniques, but are still limited to the first 12 months post transplantation. Long-term survival remains almost unchanged indicating the need to identify and improve relevant factors. Evidence in other chronically-ill patient populations shows that the healthcare system (e.g. level of chronic illness management (CIM)) and patient self-management (e.g. adherence) drive improvements in outcomes.

The BRIGHT study is the first multi-centre, multi-continental study examining healthcare system and heart transplant centres chronic illness management practice patterns and potential correlates of immunosuppressive medication nonadherence.

The knowledge gained will inform clinicians, researchers and healthcare policy makers about the level(s) interventions need to be implemented at to improve long-term outcomes for transplant recipients.

DETAILED DESCRIPTION:
Background: After receiving a heart transplant (HTx) patients have to adhere to a number of health behaviors (e.g., medication taking, and smoking cessation) in order to guarantee optimal outcomes. Non-adherence to these health behaviors is associated with poor clinical and economic outcomes. However, the prevalence of non-adherence to these health behaviors is high among HTx recipients. Furthermore, differences in prevalences among countries and continents are observed. The extent to which a HTx recipient is adherent is affected by a variety of risk factors, namely 1) patient-related factors, 2) socioeconomic factors, 3) therapy-related factors, 4) health-related factors and 5) healthcare system and team factors. To-date, this last group of factors only received limited attention in understanding the complex phenomena of adherence.

Aims: The aims of this study are:

1. To describe CIM practice patterns among centres, countries/continents in HTx.
2. To assess the prevalence and variability of nonadherence to treatment regimen, i.e. medication taking, smoking cessation, diet keeping, alcohol consumption, physical activity, sun protection and appointment keeping in HTx recipients among centres, countries/continents.
3. To determine which multi-level factors are related to immunosuppressive medication adherence at the different system levels
4. To benchmark the participating centres, countries and continents in relation to CIM practice patterns and non-adherence to health behaviours

Methodology: The BRIGHT study is an international, multi-center, cross-sectional study. Data were collected using interviews and questionnaires. HTx recipients, nurses working in the post-transplantation care of HTx recipients and the medical directors of the HTx programs were surveyed. The investigators recruited a convenience sample of 36 heart transplantation centers (North America (n= 12), European (n= 19), Australia (n= 2) and South America (n= 3)). Within participating centers, a random sample of patients who met the study eligibility criteria was selected. Per center, a minimum of 20 and a maximum of 60 patients were included. In total, 1677 heart transplant recipients were invited to participate in this study. The questionnaires used in this study will be existing questionnaires (e.g. BAASIS interview to assess adherence with medications, DASS to assess depression) as well as questionnaires developed for this study.

During a regular follow-up visit, patients were invited by a staff person to participate in this study. The staff first informed the patient about the study and, if the patient was willing to participate, retrieved a signed informed consent. Participating in this study was voluntary. Informed consent of the nurses and the medical director of the transplant center were implied by completing the questionnaires. Participant names will be held in strict confidence and will remain anonymous in research reports or publications.

The results of the benchmarking of the parameters assessed in this study will be reported by figures and tables. Because of privacy, the HTx centers can only identify the parameters specific to their center. All other information will be reported anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant patients
* 18 years or older at time of inclusion
* Transplanted and followed-up for routine care in a participating transplant center
* First transplant
* Single-organ transplant
* Between 1 and 5 years post-transplant
* Ability to read, understand and sign written informed consent (in Dutch, English, French, German, Spanish, Italian, or Portuguese, depending on the languages spoken within the country where the participating transplant center is located)
* Provided written informed consent

Exclusion Criteria:

* Receiving professional support in medication taking
* Involved in adherence-intervention research or drug trials during the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult heart transplant recipients
Sampling Method: Probability Sample
Enrollment: 1365 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported non-adherence to immunosuppressive medication | Once
  Participants will be asked about immunosuppressive medication taking during the prior 4 weeks

SECONDARY OUTCOMES:
Self-reported non-adherence to other medications (excl. immunosuppressive medications) | Once
  Participants will be asked about adherence to other medications (excl. immunosuppressive medications) during the prior 4 weeks
Self-reported adherence to smoking cessation | Once
  Participants will be asked about current and past smoking
Self-reported adherence to dietary modifications | once
  Participants will be asked about adherence to dietary recommendations during the past year
Self-reported alcohol use | Once
  Participants are asked about alcohol intake during the past year
Self-reported adherence to physical activity | Once
  Participants are asked about their level of physical activity during the past week
Self-reported adherence to sun protection | Once
  Participants will be asked about the routine use of sun protection measures
Self-reported adherence to appointment keeping | Once
  Participants will be asked if they kept the last five appointments with the transplant team

CONTACTS AND LOCATIONS:
Overall Officials: Sabina M De Geest, PhD, RN, Principal Investigator — University of Basel
Locations (1):
- University Hospitals of Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berben L, Russell C, Engberg S, Dobbels F, De Geest S. Development, content validity and inter-rater reliability testing of the Chronic Illness Management Implementation - Building Research Initiative Group: Chronic Illness Management and Adherence in Transplantation: An instrument to assess the level of chronic illness management implemented in solid organ transplant programmes. International Journal of Care Coordination. 2014;17(1-2):59-71.
- [Background] Berben L, Denhaerynck K, Dobbels F, Engberg S, Vanhaecke J, Crespo-Leiro MG, Russell CL, De Geest S; BRIGHT study consortium. Building research initiative group: chronic illness management and adherence in transplantation (BRIGHT) study: study protocol. J Adv Nurs. 2015 Mar;71(3):642-54. doi: 10.1111/jan.12519. Epub 2014 Sep 26. PMID 25257974
- [Result] Cajita MI, Denhaerynck K, Dobbels F, Berben L, Russell CL, Davidson PM, De Geest S; BRIGHT study team. Health literacy in heart transplantation: Prevalence, correlates and associations with health behaviors-Findings from the international BRIGHT study. J Heart Lung Transplant. 2017 Mar;36(3):272-279. doi: 10.1016/j.healun.2016.08.024. Epub 2016 Sep 13. PMID 27773449
- [Result] Cajita MI, Baumgartner E, Berben L, Denhaerynck K, Helmy R, Schonfeld S, Berger G, Vetter C, Dobbels F, Russell CL, De Geest S; BRIGHT Study Team. Heart transplant centers with multidisciplinary team show a higher level of chronic illness management - Findings from the International BRIGHT Study. Heart Lung. 2017 Sep-Oct;46(5):351-356. doi: 10.1016/j.hrtlng.2017.05.006. Epub 2017 Jun 16. PMID 28624338
- [Result] Senft Y, Kirsch M, Denhaerynck K, Dobbels F, Helmy R, Russell CL, Berben L, De Geest S; BRIGHT study team. Practice patterns to improve pre and post-transplant medication adherence in heart transplant centres: a secondary data analysis of the international BRIGHT study. Eur J Cardiovasc Nurs. 2018 Apr 1;17(4):356-367. doi: 10.1177/1474515117747577. Epub 2017 Dec 1. PMID 29231747
- [Result] Denhaerynck K, Berben L, Dobbels F, Russell CL, Crespo-Leiro MG, Poncelet AJ, De Geest S; BRIGHT study team. Multilevel factors are associated with immunosuppressant nonadherence in heart transplant recipients: The international BRIGHT study. Am J Transplant. 2018 Jun;18(6):1447-1460. doi: 10.1111/ajt.14611. Epub 2018 Jan 16. PMID 29205855
- [Derived] Mielke J, Cajita MI, Denhaerynck K, Valenta S, Dobbels F, Russell CL, De Geest S; BRIGHT study team. Trust in the Transplant Team Associated With the Level of Chronic Illness Management-A Secondary Data Analysis of the International BRIGHT Study. Transpl Int. 2024 Mar 11;37:11704. doi: 10.3389/ti.2024.11704. eCollection 2024. PMID 38529215
- [Derived] Rose Epstein F, Trammell J, Liu CM, Denhaerynck K, Dobbels F, Russell C, De Geest S. A Secondary Analysis from The International BRIGHT Study For Gender Differences In Adherence To Nonpharmacological Health-Related Behaviors After Heart Transplantation. Prog Transplant. 2022 Jun;32(2):138-147. doi: 10.1177/15269248221087435. Epub 2022 Mar 25. No abstract available. PMID 35331039
- [Derived] Iglesias K, De Geest S, Berben L, Dobbels F, Denhaerynk K, Russell LC, Helmy R, Peytremann-Bridevaux I; BRIGHT study team. Validation of the patient assessment of chronic illness care (PACIC) short form scale in heart transplant recipients: the international cross-sectional bright study. BMC Health Serv Res. 2020 Mar 3;20(1):160. doi: 10.1186/s12913-020-5003-3. PMID 32126998
- [Derived] Helmy R, Scalso de Almeida S, Denhaerynck K, Berben L, Dobbels F, Russell CL, de Aguiar Roza B, De Geest S; BRIGHT study team. Prevalence of Medication Nonadherence to Co-medication Compared to Immunosuppressants in Heart Transplant Recipients: Findings From the International Cross-sectional BRIGHT Study. Clin Ther. 2019 Jan;41(1):130-136. doi: 10.1016/j.clinthera.2018.11.007. Epub 2018 Dec 24. PMID 30591285
- [Derived] Helmy R, Duerinckx N, De Geest S, Denhaerynck K, Berben L, Russell CL, Van Cleemput J, Crespo-Leiro MG, Dobbels F; BRIGHT study team. The international prevalence and variability of nonadherence to the nonpharmacologic treatment regimen after heart transplantation: Findings from the cross-sectional BRIGHT study. Clin Transplant. 2018 Jul;32(7):e13280. doi: 10.1111/ctr.13280. Epub 2018 Jun 21. PMID 29754400